CLINICAL TRIAL: NCT01204229
Title: Motivational and Cognitive Intervention for College Drinkers
Acronym: MCID
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Cincinnati (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Giao Q. Tran, Ph.D., University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R21AA1AA017291A1; R21AA1AA017291A1 (Other Grant/Funding Number: R21AA1AA017291A1)
Record Dates: First submitted 2010-09-15; First posted 2010-09-17 (Estimated); Last update posted 2011-04-22 (Estimated); Status verified 2011-04

CONDITIONS: Alcohol Consumption; Anxiety; Depression
Keywords: Alcohol Consumption; Social Anxiety; Depression; Brief Intervention; Motivational Interviewing; Cognitive Behavioral Therapy; Sub-Clinical Social Anxiety; Sub-Clinical Depression
MeSH Terms: conditions — Alcohol Drinking; Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MCID (Experimental)
  Interventions: Behavioral: Motivational and Cognitive Intervention for Drinkers (MCID)
- BMI (Experimental)
  Interventions: Behavioral: Brief Motivational Intervention (BMI)

INTERVENTIONS:
Behavioral: Motivational and Cognitive Intervention for Drinkers (MCID) — Integrate social anxiety/ depression and drinking intervention
  Arms: MCID
Behavioral: Brief Motivational Intervention (BMI) — Integrate drinking intervention
  Arms: BMI

SUMMARY:
In the proposed project the investigators will develop and test a novel brief intervention targeting college students who drink heavily to cope with anxiety and depression, a behavior that increases risk for the development of alcohol dependence.

ELIGIBILITY:
Inclusion Criteria:

- 1. At least 1 heavy drinking episode (4 or more drinks for women; 5 or more drinks for men).

2. Sub-clinical anxiety or depression 3. Occasional to frequent drinking related problems

Exclusion Criteria:

* 1. Clinical Axis I diagnosis 2. Current suicidal ideation, pregnancy, major medical illness, severe alcohol dependence, current hallucinations

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-05; Primary Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
Alcohol Consumption and Drinking-Related Negative Consequences | Pre-Treatment, 2-month follow-up, 4-month follow-up, 6-month follow-up
Anxiety | Pre-Treatment, 2-month follow-up, 4-month follow-up, 6-month follow-up
Depression | Pre-Treatment, 2-month follow-up, 4-month follow-up, 6-month follow-up

SECONDARY OUTCOMES:
Cost efficacy data | 2-3 months post completion

CONTACTS AND LOCATIONS:
Overall Officials: Giao Q. Tran, Ph.D., Principal Investigator — University of Cincinnati
Locations (1):
- Psychology Department, University of Cincinnati, Cincinnati, Ohio, United States